CLINICAL TRIAL: NCT06153095
Title: A Phase 1/2 Open-label Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Efficacy of IMPT-514 in Participants With Active, Refractory Lupus Nephritis and Systemic Lupus Erythematosus
Brief Title: A Study of IMPT-514 in Active Refractory Lupus Nephritis (LN) and Systemic Lupus Erythematosus (SLE)
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Lyell Immunopharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MPCT-021N
Record Dates: First submitted 2023-11-22; First posted 2023-12-01 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2024-05

CONDITIONS: Systemic Lupus Erythematosus; Lupus Nephritis
Keywords: CAR T-cell; CD19/20; CD19; CD20; Lupus Nephritis; LN; Systemic Lupus Erythematosus; SLE; Active refractory systemic lupus erythematosus; Active refractory Lupus Nephritis
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Lupus Nephritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Phase 1 Lupus Nephritis (Experimental): Administration of IMPT-514
  Interventions: Biological: IMPT-514
- Phase 2 Lupus Nephritis (Experimental): Administration of IMPT-514
  Interventions: Biological: IMPT-514
- Phase 2 SLE without Lupus Nephritis (Experimental): Administration of IMPT-514
  Interventions: Biological: IMPT-514

INTERVENTIONS:
Biological: IMPT-514 — CAR T-cell therapy administered intravenously after a lymphodepleting therapy regimen consisting of fludarabine and cyclophosphamide
  Arms: Phase 1 Lupus Nephritis
Biological: IMPT-514 — CAR T-cell therapy administered intravenously after a lymphodepleting therapy regimen consisting of fludarabine and cyclophosphamide
  Arms: Phase 2 Lupus Nephritis
Biological: IMPT-514 — CAR T-cell therapy administered intravenously after a lymphodepleting therapy regimen consisting of fludarabine and cyclophosphamide
  Arms: Phase 2 SLE without Lupus Nephritis

SUMMARY:
This is a Phase 1/2, multi-center, open-label study evaluating the safety and efficacy of IMPT-514, a bispecific chimeric antigen receptor (CAR) targeting cluster of differentiation (CD)19 and CD20 in participants with active, refractory lupus nephritis and systemic lupus erythematosus.

IMPT-514 treatment consists of a single infusion of CAR-transduced autologous T cells administered intravenously after a lymphodepleting therapy regimen consisting of fludarabine and cyclophosphamide. Individual participants will remain in the active post-treatment period for approximately 1 year.

Participants will continue in long-term follow-up for 15 years from treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent
2. Age 18 years of age or older
3. Weight > 45 kg at enrollment
4. Adequate blood pressure control
5. On stable background therapy for autoimmune disease (LN, SLE) with stable dose of autoimmune disease medications for at least 4 weeks prior to screening
6. Diagnosis of SLE by 2019 European League Against Rheumatism (EULAR)/American College of Rheumatology (ACR) classification criteria or 2012 Systemic Lupus Collaborating Clinics (SLICC) criteria, including positive ANA or positive anti-dsDNA
7. Positive anti-nuclear antibody (ANA), anti-dsDNA (double stranded DNA) or anti-Smith antibody at screening
8. SLE participants: SLEDAI-2K ≥ 6 points, with at least 4 points on clinical, non-laboratory items
9. SLE participants: British Isles Lupus Assessment Group (BILAG) 2004 level B in 2 or more organ systems, or BILAG level A in 1 or more organ system
10. Physician Global assessment ≥ 1 on 0 to 3 visual analogue scale (VAS)
11. LN participants: Active, biopsy-proven, proliferative LN Class III or IV by 2018 International Society of Nephrology/Renal Pathology Society (ISN/RPS) criteria

Other protocol-defined criteria apply.

Exclusion criteria:

1. Any clinically significant underlying illness, other than SLE and LN, which would pose a safety risk or concern, as determined by the Investigator
2. Any other systemic autoimmune condition
3. Rapidly progressive glomerulonephritis
4. Active central nervous system (CNS) lupus
5. History of allogeneic bone marrow or stem cell transplantation or solid organ transplantation
6. History of prior B cell directed cell therapy, including CAR T treatment, autologous or allogeneic, as well as prior bispecific or T cell engager therapy
7. Drug-induced SLE

Other protocol-defined criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2025-01-09 (Actual); Study Completion 2025-01-09 (Actual)

PRIMARY OUTCOMES:
Phase I: Incidence of dose limiting toxicities (DLTs), serious adverse events (SAEs), and other treatment-emergent adverse events (TEAEs). | Baseline to Month 6
Phase I: Incidence of TEAEs, percent reduction in peripheral B cells, and the proportion of enrolled participants who receive the target dose. | Baseline to Month 6
Phase II: Cohort 1 (LN): Proportion of participants with Complete Renal Response (CRR) as defined by EULAR/ERA-EDTA at Month 6. | Baseline to Month 6
Phase II: Cohort 2 (SLE): Proportion of participants achieving definition of remission in SLE (DORIS) at Month 6. | Baseline to Month 6

CONTACTS AND LOCATIONS:
Locations (4):
- United States (3):
  - University of California, Los Angeles (UCLA) Medical Center, Los Angeles, California
  - University of California San Francisco, San Francisco, California
  - University of Iowa, Iowa City, Iowa
- Westmead Hospital, Westmead, Australia

IPD SHARING:
Plan to Share IPD: No